CLINICAL TRIAL: NCT02849873
Title: Randomized Study Evaluating the Absorption and Systematic Pharmacokinetics of Topically Applied IDP-123 Lotion in Comparison With Tazorac Cream in Subjects With Moderate to Severe Acne Vulgaris Under Maximal Use Conditions
Brief Title: Absorption and Systematic Pharmacokinetics of IDP-123 Lotion in Comparison With Tazorac Cream
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V01-123A-501
Record Dates: First submitted 2016-07-06; First posted 2016-07-29 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — tazarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IDp-123 Lotion (Experimental): Lotion
  Interventions: Drug: IDP-123 Lotion
- Tazorac Cream (Active Comparator): Cream
  Interventions: Drug: Tazorac Cream

INTERVENTIONS:
Drug: IDP-123 Lotion — Lotion
  Other Names: IDP-123
  Arms: IDp-123 Lotion
Drug: Tazorac Cream — Cream
  Other Names: Tazorac
  Arms: Tazorac Cream

SUMMARY:
The Absorption and Systematic Pharmacokinetics of IDP-123 Lotion in Comparison with Tazorac Cream.

DETAILED DESCRIPTION:
Randomized study evaluating the absorption and systematic pharmacokinetics of IDP-123 lotion in comparison with Tazorac Cream in subjects with moderate to severe acne vulgaris under maximal use conditions.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female, at least 9 years of age (at least 12 years of age for Tazorac Cream).
* Verbal and written informed consent must be obtained. Subjects less than age of consent must sign an assent for the study and a parent or a legal guardian must sign the informed consent (if the subject reaches age of consent during the study they should be re-consented at the next study visit).
* Subject must have a score of 3 (moderate) or 4 (severe) on the Evaluator's Global Severity assessment at the screening and baseline visit.
* Subjects with facial acne inflammatory lesion count no less than 20 but no more than 40.
* Subjects with facial acne non-inflammatory lesions count no less than 20 but no more than 100.

Key Exclusion Criteria:

* Use of an investigational drug or device within 30 days of enrollment or participation in a research study concurrent with this study.
* Any dermatological conditions on the face that could interfere with clinical evaluations such as acne conglobate, acne fulminans, secondary acne, perioral dermatitis, clinically significant rosacea, gram-negative folliculitis, dermatitis, eczema.
* Any underlying disease or some other dermatological condition of the face that requires the use of interfering topical or systemic therapy or makes evaluations and lesion count inconclusive.
* Subjects with a facial beard or mustache that could interfere with the study assessments.
* Subjects with more than 2 facial nodules.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Evaluator's Global Severity Score: At Day 15 (or ET), acne severity will be determined by the investigator/evaluator based on a global assessment of the inflammatory and non-inflammatory lesions of facial acne. | 15 Days
  Evaluations will be graded on a static scale ranging from 0 (clear) to 4 (severe)

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, Study Director — Valeant Pharmaceuticals
Locations (1):
- Valeant Site 01, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes